CLINICAL TRIAL: NCT00827502
Title: Trulimax (Azithromycin ) Non-Interventional Study In Acute Bacterial Upper Respiratory Tract Infections
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A0661198
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Upper Respiratory Tract Infections
Keywords: TRULIMAX (AZITHROMYCIN ) NON-INTERVENTIONAL STUDY
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess effectiveness of Trulimax (Azithromycin) in Acute Bacterial Upper Respiratory Tract Infections (URTIs).

DETAILED DESCRIPTION:
Prospective, Open-label, Non-interventional and Multi-center Study NA

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Patients with acute URTI, presumed to be of bacterial origin as per the clinical judgment of the investigator.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only patients with acute URTI, presumed to be of bacterial origin as per the clinical judgment of the investigator will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- India (9):
  - Pfizer Investigational Site, Jn Vishakhapatnam, Andhra Pradesh
  - Pfizer Investigational Site, Visakhapatnam, Andhra Pradesh
  - Pfizer Investigational Site, Guwhati, Assam
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Vāshi, Maharashtra
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Delhi, New Delhi
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661198&StudyName=Trulimax%20%28Azithromycin%20%29%20Non-Interventional%20Study%20In%20Acute%20Bacterial%20Upper%20Respiratory%20Tract%20Infections

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: The use and dosage recommendations for Azithromycin took place on the basis of the approved local product document (LPD) and were adjusted solely according to medical and therapeutic necessities. According to the approved LPD, in general a total dose of 30 mg/kg was given as a single daily dose(10 mg/kg daily for 3 days, or given over 5 days with a single daily dose of 10 mg/kg on day 1, and then reduced to 5 mg/kg on days 2 to 5). For children with acute otitis media a single dose of 30 mg/kg was recommended. Children with streptococcal pharyngitis were given a single dose of 10 mg/kg or 20 mg/kg for 3 days and did not exceed a daily dose of 500mg. The maximum recommended total dose of Azithromycin in children for any treatment was 1500 mg. Azithromycin tablets were administered only to children weighing more than 45 kg.
Period: Overall Study
Arm/Group | Azithromycin
Started | 421
Received Treatment (Number Treated) | 410
Completed | 400
Not Completed | 21
Not completed — randomized but not treated | 11
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin
Number analyzed (Participants) | 410
Age, Customized [Number; unit: participants]
  <18 years | 51
  18-44 years | 270
  45-64 years | 73
  >= 65 years | 9
  Unspecified | 2
  Demographic information not collected | 5
Sex/Gender, Customized [Number; unit: participants]
  Female | 155
  Male | 245
  Unspecified | 5
  Demographic information not collected | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Investigator Assessment of Clinical Outcome (Success/Failure) at End of Study
Description: Success: Cure (disappearance of all pre-treatment signs and symptoms of infection) or improvement in or partial disappearance of signs and symptoms not requiring further treatment at end of study; Failure: No change in, or worsening of baseline signs and symptoms requiring modification of treatment, ie, addition of or switch to another systemic antibacterial therapy. Unknown or missing values were considered as failure.
Time Frame: Baseline to 2 weeks
Population: The full analysis set (FAS) included all subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 408
participants
  Success | 275
  Failure (Unknown or missing values also included) | 133

2. Secondary Outcome: Cost (in Indian Rupees) Per Participant of Utilizations Including General Consultations, Medications, Chest X-ray, Complete Blood Count, and Erythrocyte Sedimentation Rate
Description: Cost (in Indian Rupees) per participant of utilizations including general consultations over the study; each medication over the study (study drug, analgesics, antipyretics, anti-inflammatory drugs, vitamins, other study medication), radiological tests over the study (chest X-ray); and clinical laboratory tests over the study (complete blood count and erythrocyte sedimentation rate).
Time Frame: Baseline to 3 months
Population: FAS
Measure: Median (Full Range); unit: cost (in Indian Rupees) per participant
Arm/Group | Azithromycin
Number analyzed (Participants) | 410
cost (in Indian Rupees) per participant
  General Consultations (n=346) | 500 [150 to 1300]
  Overall Study Drugs (n=390) | 170 [85 to 272]
  Analgesics (n=205) | 18 [2 to 112]
  Antipyretics (n=116) | 9 [1 to 21]
  Anti-inflammatory (n=88) | 20 [2 to 84]
  Vitamins (n=180) | 20 [2 to 70]
  Other study medication (n=235) | 20 [2 to 96]
  Chest X-ray (n=9) | 150 [150 to 150]
  Complete Blood Count (n=15) | 200 [200 to 200]
  Erythrocyte Sedimentation Rate (n=4) | 80 [80 to 80]

3. Primary Outcome: Number of Subjects With an Investigator Assessment of Clinical Outcome (Cure/Improvement/Failure) at End of Study
Description: Cure: Disappearance of all pre-treatment signs and symptoms of infection; Improvement: Improvement in, or partial disappearance of signs and symptoms without requiring further antibacterial therapy. Subjects who discontinued study drug for reasons other than lack of clinical response, i.e., despite clinical improvement, were included in this category; and Failure: No change in, or worsening of baseline signs and symptoms requiring modification of treatment, ie, addition of or switch to another systemic antibacterial therapy. An unknown response or missing value was considered clinical failure.
Time Frame: Baseline to 2 weeks
Population: The efficacy evaluable (EVAL) population included subjects in the FAS having at least 1 definitive follow up global response assessment to treatment of URTIs.
Measure: Number; unit: Participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 278
Participants
  Cure | 249
  Improvement | 26
  Failure | 3

ADVERSE EVENTS:
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/410
Other Adverse Events (participants affected / at risk) | 16/410
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=410)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastric disorder (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Adverse event (General disorders) | 1
Drug intolerance (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.